CLINICAL TRIAL: NCT06668649
Title: Validation of Polish Language Version of Fatigue Severity Scale
Brief Title: Polish Version Fatigue Severity Scale
Status: Recruiting | Type: Observational
Sponsor: Jakub Antczak (Other)
Collaborators: Institute of Psychiatry and Neurology, Warsaw (Other)
Responsible Party: Sponsor-Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Organization: Jagiellonian University (Other)
Other Study IDs: JagiellonianU74
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Amyotrophic Lateral Sclerosis; Stroke, Ischemic
Keywords: Fatigue; Multiple Sclerosis; stroke; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Amyotrophic Lateral Sclerosis; Ischemic Stroke; Fatigue; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Both sexes, aged 18 or older. The group will include 80 patients with multiple sclerosis, 80 patients with amyotrophic lateral sclerosis and 50 survivors of ischemic stroke
  Interventions: Diagnostic Test: Testing with Questionnaires
- Control: Both sexes, aged 18 or older. The group will include 100 healthy controls.
  Interventions: Diagnostic Test: Testing with Questionnaires

INTERVENTIONS:
Diagnostic Test: Testing with Questionnaires — Testing with following Questionnaires: pFSS, Polish-language version of Modified Fatigue Impact Scale, Visual Analogue Scale of Fatigue, EQ-5D-5L (EuroQol-5 dimension) questionnaire, Beck Depression Inventory II. In randomly selected 30 patients and 20 controls questionnaires will be administered twice with two weeks interval to assess the test-retest reliability.

SUMMARY:
Fatigue is one of main symptoms in multiple sclerosis, amyotrophic lateral sclerosis and other diseases with profound effect on quality of life and professional and social functioning. Not infrequent it is misdiagnosed as sleepiness or other symptom. Fatigue severity scale is a time efficient and easy to apply instrument to assess the impact of fatigue on patient's life. The aim of this study is to validate the Polish-language version of the Fatigue Severity Scale.

DETAILED DESCRIPTION:
Fatigue is one of main symptoms in multiple sclerosis, amyotrophic lateral sclerosis, post-polio syndrome, stroke, parkinsonism as well as in the chronic fatigue syndrome. It has profound effect on quality of life and professional and social functioning and in multiple sclerosis it is described as the worst symptoms by the 50% of patients. It is defined as the difficulty in initiating and maintaining a sustained mental or physical activity. Not infrequent it is misdiagnosed as sleepiness or other symptom. Fatigue severity scale (FSS) is a time efficient and easy to apply instrument to assess the impact of fatigue on patient's life. It has been translated and validated in Turkish, Russian, Hindi, Portuguese, and many other languages. FSS is a short, nine-item self-report questionnaire. Each item is a Likert scale, scored from one to seven, where seven refers to the most severely expressed aspect of fatigue. The aim of this study is to validate the Polish-language version of the Fatigue Severity Scale (pFSS). This version has been created according to widely accepted, respective standards, including translation by two independent native Polish-language speakers with acquired knowledge of English and backward translation by two independent native English-language speakers with acquired knowledge of Polish as well as with the pretesting on ten patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite multiple sclerosis or definite, laboratory-supported multiple sclerosis, or definite amyotrophic lateral sclerosis, or probable amyotrophic lateral sclerosis or probable, laboratory supported amyotrophic lateral sclerosis or ischemic stroke or - for healthy controls - lack of diseases, pharmacotherapy or habits, which could induce abnormal tiredness

Exclusion Criteria:

* Presence of cognitive deficits or behavioral disorder, which could disturb participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the neurologic ambulatories and neurologic clinics of Jagiellonian University Medical College in Cracow and of Institute of Psychiatry and Neurology in Warsaw. Healthy controls will be recruited from personel of those facitlites as well as from the relatives of members of research team.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Internal Consistency | Through study completion, an average of 1 year
  Consistency between particular items of Polish language version of the Fatigue Severity Scale will be evaluated using Cronbach alfa test. The score of the Polish language version of the Fatigue Severity Scale ranges between 9 and 63 with higher scores meaning a worse outcome.
Validity | Through study completion, an average of 1 year
  Validity will be tested by calculating the correlation of Polish language version of the Fatigue Severity Scale score with scores of Polish-language version of Modified Fatigue Impact Scale. The score of the Polish language version of the Fatigue Severity Scale ranges between 9 and 63 with higher scores meaning a worse outcome. The score of the Modified Fatigue Impact Scale ranges between 0 and 84 with higher scores meaning a worse outcome.
Reliability | Through study completion, an average of 1 year
  Reliability will be tested by calculating the correlation between Polish language version of the Fatigue Severity Scale scores from the 1st and 2nd administration in the randomly selected subgroup of patients and controls. The score of the Polish language version of the Fatigue Severity Scale ranges between 9 and 63 with higher scores meaning a worse outcome.

SECONDARY OUTCOMES:
Impact of fatigue on quality of life - index | Through study completion, an average of 1 year
  Correlation between Polish language version of the Fatigue Severity Scale score and the index score of EQ-5D-5L (EuroQol-5 dimension) questionnaire. The score of the Polish language version of the Fatigue Severity Scale ranges between 9 and 63 with higher scores meaning a worse outcome. The index score of EQ-5D-5L (EuroQol-5 dimension) questionnaire ranges between -0.59 to 1 with higher scores indicating better outcome.
Impact of fatigue on quality of life - visual analogue scale | Through study completion, an average of 1 year
  Correlation between Polish language version of the Fatigue Severity Scale score and the visual analogue scale score of EQ-5D-5L (EuroQol-5 dimension) questionnaire. The score of the Polish language version of the Fatigue Severity Scale ranges between 9 and 63 with higher scores meaning a worse outcome. The visual analogue scale score of EQ-5D-5L (EuroQol-5 dimension) questionnaire ranges between 0 to 100 with higher scores indicating better outcome.
Impact of fatigue on depression | Through study completion, an average of 1 year
  Correlation between Polish language version of the Fatigue Severity Scale score and score of Beck Depression Inventory II. The score of the Polish language version of the Fatigue Severity Scale ranges between 9 and 63 with higher scores meaning a worse outcome. The score of the Beck Depression Inventory II ranges between 0 and 63 with higher scores indicating worse outcome.
Difference in fatigue level between patients and controls | Through study completion, an average of 1 year
  Difference in Polish language version of the Fatigue Severity Scale score between patients and controls. The score of the Polish language version of the Fatigue Severity Scale ranges between 9 and 63 with higher scores meaning a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub M Antczak, MD, Principal Investigator — Jagiellonian University
Locations (2):
- Poland (2):
  - Jagiellonian University Medical College, Department of Neurology, Krakow, Lesser Poland Voivodeship
  - Institute of Psychiatry and Neurology, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the scans of collected questionnaires will be available upon request sent to the e-mail: jakub.antczak@uj.edu.pl
Supporting Information: Study Protocol
Time Frame: After the study is completed for the period of ten years.
Access Criteria: Researchers affiliated in institutions listed on clinicaltrials.gov.

REFERENCES:
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569